CLINICAL TRIAL: NCT02333422
Title: Clinical Trial Using NIRS Neurofeedback on Children With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: NIRS Neurofeedback as a Treatment for Attention Deficit Hyperactivity Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-0061
Record Dates: First submitted 2014-12-30; First posted 2015-01-07 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: NIRS Neurofeedback; Attention Deficit Hyperactivity Disorder; Near Infrared Spectroscopy; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NIRS Neurofeedback (Experimental): NIRS Neurofeedback training of frontal and pre frontal lobes activation. The intervention consist of 24 NIRS neurofeedback sessions over 12 weeks, 2 sessions per week.
  Interventions: Other: NIRS Neurofeedback

INTERVENTIONS:
Other: NIRS Neurofeedback — The sensor will be placed on 4 specific regions defined by the International 10/20 System for Electrode Placement. F7, Fp1, Fp2 and F8. Each region will be initially trained for 4 minutes, with the eyes open, gradually increasing training time throughout the sessions to a maximum of 10 minutes. Training will amount to 24 sessions, occurring 2 times per week over a period of 3 moths. The procedure will be interrupted at any time, should the subject demonstrate the desire to stop.
  Other Names: Near Infrared Spectroscopy Neurofeedback

SUMMARY:
The investigators therefore propose a pilot study to establish the effectiveness of NIRS Neurofeedback training in reducing the intensity of ADHD symptom expression on children, improvement of the cognitive and global functions associated with ADHD, effects on cerebral blood perfusion in the cortex and safety plus possible unknown side-effects.

DETAILED DESCRIPTION:
Background:

Attention Deficit Hyperactivity Disorder (ADHD) is a mental condition originating in childhood, characterized by symptoms of lack attention, hyperactivity and impulsiveness associated with significant functional impairment. Currently, the use of neurofeedback as a non-drug alternative technique for treatment of ADHD has increasingly spread among the clinical and academic fields, producing relevant findings with regard to its effectiveness. The SCP Neurofeedback and EEG Neurofeedback have been the most studied techniques until the moment, with equipments and systems made available to the market at prices between US$ 10.000 and US$ 20.000, while NIRS Neurofeedback equipments can be found for around US$ 2.000. Due to the low cost of the necessary equipment's and easy access to the technology, the use of NIRS Neurofeedback was opted for in the search to evaluate the techniques effectiveness in the improvement of ADHD symptoms as well as the patients' cognitive performance.

This research is an open label treatment trial with NIRS Neurofeedback training of frontal and pre frontal lobes activation in children school-aged 7 - 12 years old with ADHD. Ten participants will be recruited over 3 months and will be offered 24 NIRS Neurofeedback sessions over 12 weeks, 2 sessions per week. The present study will be carried out as part of the care routine of the Child and Adolescent Psychiatry Services at Hospital de Clínicas de Porto Alegre. Primary outcome will be standard clinical behavioural rating scales. Secondary outcomes will include neuropsychological parameters, neurofunctional parameters using SPECT (Single Photon Emission Computed Tomography), global function, quality of life assessment, side effects and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ADHD clinically.
* Cognitive dysfunction: ≥11/2; standard deviation above norm in at least two neuropsychological measurements: executive functions (inhibitory control), gratification aversion and time processing
* Not having used ADHD medication in at least three months with parental consent for not treating ADHD with medication

Exclusion Criteria:

* Existence of another co-morbid mental disorder which is clinically relevant and demands treatment
* IQ < 80

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Diagnostic and severity measure | 3 months
  Swanson, Nolan and Pelham Questionnaire version IV (SNAPIV)

SECONDARY OUTCOMES:
Basic processing | 3 months
  Using Two-choice Reaction Time Task
Inhibition control | 3 months
  Using Go/No-Go test
Conflict Control | 3 months
  Using Modified Stroop Task
Time processing | 3 months
  Using Time Anticipation (400ms e 2000ms)
Delay Aversion | 3 months
  Using Choice Delay Task combined with Delay Reaction Time
Cerebral blood perfusion | 3 months
  Using SPECT (Single Photon Emission Computed Tomography) toward identifying changes to cerebral blood perfusion in the trained areas (F7, Fp1, Fp2 e F8) and all cortex
Psychiatric and social function measure | 3 months
  Children's Global Assessment Scale (CGAS) is an adaptation of the Global Assessment Scale (GAS) for young people aged 4-16 years
Treatment response assessment | 3 months
  CGI (Clinical Global Impression)
Quality of life | 3 months
  Quality of life evaluation scale (AUQEI)
Side Effects | 3 months
  Using SERS (Barkley's Side Effect Rating Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Luis AP Rohde, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil